CLINICAL TRIAL: NCT06329804
Title: The Dose Response Effect of Isometric Handgrip Training Frequency on Blood Pressure: a Randomised Controlled Trial in Normotensive Individuals
Brief Title: The Dose Response Effect of Isometric Handgrip Training Frequency on Blood Pressure in Normotensive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Collaborators: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RM_01-11-21b
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-03

CONDITIONS: Blood Pressure
Keywords: Blood Pressure; Isometric Handgrip Exercise; Dose Response; Training Frequency; Perceptual Responses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Intervention Control (No Intervention): Participants allocated to this group will maintain their usual lifestyle for 4-weeks
- Two Sessions/Week (Experimental): Participants allocated to this group will complete 4-weeks of isometric handgrip exercise training with a frequency of two sessions/week
  Interventions: Other: Isometric Handgrip Exercise Training (IHGT)
- Four Sessions/Week (Active Comparator): Participants allocated to this group will complete 4-weeks of isometric handgrip exercise training with a frequency of four sessions/week
  Interventions: Other: Isometric Handgrip Exercise Training (IHGT)

INTERVENTIONS:
Other: Isometric Handgrip Exercise Training (IHGT) — Each IHGT session will consist of 4 x 2-minute contractions at 30% maximal voluntary contraction, with 2-minutes of rest in between, performed with the dominant hand. Training will be performed using an electronic hand dynamometer (Camry EH101, Zhongshan Camry Electronic Co. Ltd, Guangdong).
  Arms: Four Sessions/Week; Two Sessions/Week

SUMMARY:
It is estimated by WHO (2021) that 1.4 billion individuals across the globe have high blood pressure with only 14% of people managing these elevated levels. Simple and effective lifestyle strategies are required to help people improve their blood pressure and/or attenuate increases in blood pressure with ageing. Exercise is one possible strategy: in previous research, several different types of exercise have been shown to have effects on blood pressure (Blackwell et al., 2017). However, many individuals do not adhere to currently recommended levels of exercise (150 mins of moderate intensity exercise per week), due to a combination of the required time commitment, lack of motivation, and the associated levels of effort / exertion and discomfort (Korkiakangas et al 2009). Thus, there is a need to investigate alternative exercise interventions which will overcome these barriers but remain effective at improving blood pressure (Herrod, Lund, & Phillips, 2021).

Low intensity isometric hand grip training (IHGT) has been shown to result in large decreases in rest-ing blood pressure in younger and older age groups, in both men and women, and in individuals with normal as well as elevated baseline blood pressure (Badrov et al, 2013; Bentley et al., 2018; Millar et al., 2014). In this research, IHGT has typically involved performing 4 x 2 IHGT holds at 30% of maximal voluntary contraction, 3 times a week, over a 4-8-week intervention (Millar et al, 2014). Interestingly, there are very few studies that have investigated the effect of changing different protocol parameters on the adaptations in blood pressure, and the minimal effective dose of IHGT is unknown. One important modifiable parameter is training frequency and it is unknown whether reducing the frequency of IHGT will reduce the efficacy for improving blood pressure. Therefore, the aim of this randomised controlled trial is to compare the effect of IHGT with a frequency of 2 or 4 sessions/week on resting blood pressure.

DETAILED DESCRIPTION:
Data collection for this study will take place at two University sites: Swansea University in The UK and National Taiwan Normal University in Taiwan. Separate ethical approval will be sought at each site.

Participants

The primary outcome in this study will be the change in clinic measured systolic blood pressure. In a meta-analysis of 147 RCTs, a 10 mmHg decrease in SBP reduced CHD events by 22% (Law 2009). We powered this study to be able to detect a smallest worthwhile effect of 3.0 mmHg (equivalent to a CHD risk reduction of ~7%). Based on the standard deviation of repeated measures of systolic blood pressure of ~2.9 mmHg in our laboratory, a sample size of 45 participants (15 per group) will achieve 80% power to detect this difference with an alpha of 0.05. Therefore, in order to ensure equal recruitment across both study sites, we will recruit up 30 participants (10 per group) at each site. Participants will be low active men and women who do not currently meet the recommended physical activity guidelines (age range: 18-40 years).

The study protocol will be fully explained to all subjects in written and verbal form before they are asked to provide written consent. Participants will be randomised to one of three experimental groups, performing either 2 or 4 isometric handgrip training sessions per week for 4 weeks, or a no-intervention control.

Baseline Testing

Participants will be asked to attend the sport and exercise science laboratory at Swansea University Bay Campus for a baseline assessment of blood pressure. Participants will be asked to refrain from any strenuous exercise for 2 days prior and from consuming any alcohol for 1 day prior to testing. Caffeine intake will be permitted in the day prior to testing but we will ask participants to complete a 1-day food diary (including caffeine containing products) prior to the baseline testing and we will ask participants to replicate this diet prior to the post-training assessment. Participants will attend the lab in the morning between 8 and 10am after fasting (water only) from 10pm the previous even-ing. To ensure they are hydrated they will be asked to consume 1 pint of water immediately upon waking.

Participants' blood pressure will be measured following a 10-minute rest period in a supine position in a dark room. Blood pressure will then be measured in the (unclothed) left arm using an automat-ed monitor (Omron MIT elite plus) whilst participants remain in the supine position. Blood pressure will be measured three times with 1 minute rest intervals in between. If there is a less than 5 mmHg difference between the final two readings, then the mean of these two readings will be taken forward for analysis (Pickering et al, 2005). If there is a difference >5 mmHg between the two readings, then 2 additional readings will be taken and the mean of the 4 readings will be taken for-ward for analysis (Pickering et al, 2005). Arm circumference will be measured prior to the blood pressure measurement to determine the correct cuff size.

Following blood pressure assessment, participants will be randomised to their experimental group using the envelope method. Participants who are randomised to the IHGT group will be asked to perform a 1 repetition maximum for an isometric handgrip contraction, to determine IHGT intensity. The best of 3 measurements of the dominant arm will be used to determine training intensity.

IHGT intervention

Participants allocated to the IHGT groups will complete a 4-week home-based IHGT intervention involving either 2 or 4 sessions per week. Each session will consist of 4 x 2-minute contractions at 30% maximal voluntary contraction, with 2-minutes of rest in between, performed with the dominant hand. Training will be performed using an electronic hand dynamometer (Camry EH101, Zhongshan Camry Electronic Co. Ltd, Guangdong).

Training sessions will be scheduled on weekdays and all sessions will be supervised by 1 member of the research team via Zoom to ensure compliance and training fidelity. During every session, the researcher will record the contraction tension every 15 seconds during each 2-minute contraction. In addition, during the first session of each training week, a rating of perceived exertion (Borg scale) and affective valence (feeling scale) will be measured every 30 seconds, during each 2-minute contraction.

Post-Training Testing

Resting blood pressure and grip strength will be measured three days following the final training session using identical procedures to the pre-training assessment (described above).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years
* Scoring 'low' on the international physical activity questionnaire (IPAQ)
* Apparently healthy with no indications of chronic disease according to a self-report health history questionnaire and the physical activity readiness questionnaire.
* Resting blood pressure <140/90 mmHg during baseline assessment.

Exclusion Criteria:

* Aged <18 or >40 years
* Previously diagnosed with hypertension and/or currently taking anti-hypertensive medication.
* Any contraindication to exercise based on responses to the self-report health-history questionnaire or the physical activity readiness questionnaire.
* Scoring moderate or high on the international physical activity questionnaire (IPAQ).
* Resting blood pressure >140/90 mmHg during baseline assessment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Resting Systolic Blood Pressure | 4 weeks
  Resting systolic blood pressure will be measured before training commences and then 3 days after the final exercise session.

SECONDARY OUTCOMES:
Resting Diastolic Blood Pressure | 4 weeks
  Resting diastolic blood pressure will be measured before training commences and then 3 days after the final exercise session.
Resting Mean Arterial Blood Pressure | 4 weeks
  Resting mean arterial blood pressure will be measured before training commences and then 3 days after the final exercise session.

OTHER OUTCOMES:
Ratings of perceived exertion | 4 Weeks (Week 1 and Week 4)
  ratings of perceived exertion will be measured during the acute isometric handgrip exercise sessions using the 6-20 Borg Scale. Measurements will be collected every 30-seconds during each two minute contraction.
Affective Valence | 4 Weeks (Week 1 and Week 4)
  Affective valence will be measured during the acute isometric handgrip exercise sessions using the Feeling Scale. Measurements will be collected every 30-seconds during each two minute contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Metcalfe, PhD, Principal Investigator — Swansea University
Locations (2):
- National Taiwan Normal University, Taipei, Taiwan
- Swansea University, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No